CLINICAL TRIAL: NCT06804486
Title: Exercise and Physical Activity in Children With Pediatric Acquired Brain Injury
Acronym: DIScover_Ped
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Andrea Gutiérrez Suárez, PhD, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: DIScover_Pediatric
Record Dates: First submitted 2025-01-23; First posted 2025-02-03 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-01

CONDITIONS: Acquired Brain Injury
Keywords: PEDIATRIC ACQUIRED BRAIN INJURY; exercise; physical-sports activity; intervention
MeSH Terms: conditions — Brain Injuries; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active PEDIATRIC ACQUIRED BRAIN INJURY (Experimental)
  Interventions: Behavioral: Exercise; Other: Recommendation to Deprescribe
- non active PEDIATRIC ACQUIRED BRAIN INJURY (No Intervention): non active PEDIATRIC ACQUIRED BRAIN INJURY

INTERVENTIONS:
Behavioral: Exercise — Exercise and physical-sports activity program
  Other Names: exercise and physical-sports activity
  Arms: active PEDIATRIC ACQUIRED BRAIN INJURY
Other: Recommendation to Deprescribe — Recommendation to Deprescribe
  Arms: active PEDIATRIC ACQUIRED BRAIN INJURY

SUMMARY:
Exercise and physical activity in children with pediatric acquired brain injury

DETAILED DESCRIPTION:
Although emerging approaches have emerged in the design of interventions that promote an orientation towards physical activity scientific evidence on their efficacy in this particular population remains limited. This underscores the need for further research to evaluate the efficacy of these intervention approaches in the context of pediatric ABI.

ELIGIBILITY:
Inclusion Criteria:

* Be under 18 years of age and present a medical diagnosis of pediatric acquired brain injury.
* Have the informed consent completed and signed
* Present a state that allows following indications for the practice of exercise and physical-sports activity.

Exclusion Criteria:

* Have medical comorbidities that contraindicate the safe performance of the program (i.e., cardiac or respiratory instability, uncontrolled seizures).
* Have additional disabling conditions, such as cognitive impairment and/or an inability to communicate with the researcher verbally, in writing, or through an emissary.
* Non-attendance and/or non-collaboration at 70% of the sessions of the program.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Through study completion, an average of 1 year
  Pediatric Quality of Life PedsQL

SECONDARY OUTCOMES:
Functionality | Through study completion, an average of 1 year
  Berg Balance Scale and Timed Up and Go

CONTACTS AND LOCATIONS:
Locations (1):
- Niño Jesus Hospital, Madrid, Madrid, Spain